CLINICAL TRIAL: NCT01577654
Title: A Randomized, Open-label Phase 2 Study of EC145 Single-agent and the Combination of EC145 Plus Docetaxel Versus Docetaxel Alone in Participants With Folate-receptor Positive [FR(++)] Second Line NSCLC
Brief Title: Phase 2 Study of EC145 Alone Versus EC145+Docetaxel Versus Docetaxel Alone in Participants With FR(++) 2nd Line Non Small Cell Lung Cancer
Acronym: TARGET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8109-003; 2012-000966-40 (EudraCT Number)
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: adenocarcinoma; squamous; adenosquamous; adenocarcinoma with other NSCLC variants; EC145; EC20; Vintafolide; Etarfolatide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma | interventions — EC145; Docetaxel; technetium 99m etarfolatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: EC145 alone (Experimental): EC145 alone
  Interventions: Drug: EC145; Drug: EC20
- Arm B: EC145 + Docetaxel (Experimental): EC145 + Docetaxel
  Interventions: Drug: EC145 + Docetaxel; Drug: EC20
- Arm C: Docetaxel alone (Active Comparator): Docetaxel alone
  Interventions: Drug: Docetaxel; Drug: EC20

INTERVENTIONS:
Drug: EC145 — 2.5 mg on Days 1,4,8,11 (Weeks 1 and 2 q3 weeks)
  Other Names: Vintafolide
  Arms: Arm A: EC145 alone
Drug: EC145 + Docetaxel — EC145 2.5 mg on Days 1,4,8,11 (Weeks 1 and 2 q3 weeks) +
  Docetaxel 75 mg/m2 IV Day 1 q 3 weeks
  Other Names: Vintafolide; Taxotere
  Arms: Arm B: EC145 + Docetaxel
Drug: Docetaxel — 75 mg/m2 IV Day 1 q 3 weeks
  Other Names: Taxotere
  Arms: Arm C: Docetaxel alone
Drug: EC20 — During the screening period participants will receive a single intravenous administration of EC20 prior to SPECT imaging
  Other Names: Etarfolatide

SUMMARY:
This study will test the activity of single-agent EC145 and the combination of EC145 plus docetaxel against the current standard docetaxel in second line Non Small Cell Lung Cancer (NSCLC) (adenocarcinoma, squamous, adenosquamous or adenocarcinoma with other NSCLC variants of the lung) in participants with all target lesions expressing the folate receptor [FR(++)].

DETAILED DESCRIPTION:
In a phase 2 study of single-agent EC145 in heavily pretreated non-small cell lung cancer (NSCLC) patients (median of 3 prior chemotherapy regimens), the subgroup with all target lesions expressing the folate receptor [FR(++)] had a promising prolonged progression free survival of 7.1 months and overall survival of 10.9 months. Furthermore, in-vitro and in-vivo studies in KB models showed good synergism between EC145 and docetaxel.

This study will clinically assess for the first time the combination of EC145+docetaxel (Arm B) in participants with NSCLC (Stage IIIB or IV). This is an international, multicenter, centrally randomized, open-label, phase 2 study comparing single-agent EC145, EC145+docetaxel combination therapy, and single-agent docetaxel in participants with NSCLC who have failed one prior chemotherapy and who have all target lesions expressing the folate receptor [FR(++)]. Eligible participants will be randomized in a 1:1:1 ratio into either Arm A (single-agent EC145), Arm B (EC145+docetaxel combination therapy), or Arm C (single-agent docetaxel) and will receive treatment until either disease progression or intolerable toxicity.

This study is intended to investigate if there is a sufficiently strong efficacy signal in order to proceed with phase 3 testing with either EC145 single-agent and/or the combination of EC145+docetaxel against the standard-of-care docetaxel in second-line NSCLC.

This study will clinically assess for the first time the combination of EC145+docetaxel (Arm B) in participants with NSCLC (Stage IIIB or IV). Therefore, an interim safety analysis will be done by the DSMB after 5 participants in Arm B have completed 1 cycle of therapy, and the second analysis after 15 participants in Arm B have completed 1 cycle of therapy.

If the majority of the enrolled participants (more than 70%) require a dose reduction of one level (to 60 mg/m2), the dose will be reduced for the remainder of the study. If the majority of the participants (more than 70%) require 2 dose reductions (to 40 mg/m2), the sponsor will consider discontinuing the combination arm.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to sign an approved informed consent form (ICF).
2. Must be ≥ 18 years of age.
3. Histology confirmed diagnosis of non-small cell lung cancer (adenocarcinoma, squamous, adenosquamous, or adenocarcinoma with other NSCLC variants of the lung) (Stage IIIB or IV).
4. All (RECIST v1.1-defined) target lesions positive for the folate receptor [FR(++)] by SPECT scan.
5. Only one prior systemic therapy for advanced disease (e.g.,a platinum doublet or a maintenance regimen that includes a platinum doublet; in addition, the participant may have received an epidermal growth factor receptor [EGFR] inhibitor).
6. Radiological evaluation conducted no more than 28 days prior to beginning study therapy. If history of CNS metastasis baseline radiological imaging must include brain MRI or CT.
7. Radiologic evidence of disease progression following the most recent prior treatment.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
9. Must have recovered (to baseline/stabilization) from prior cytotoxic-therapy-associated acute toxicities.
10. Prior radiation therapy is allowed if the following criteria is met:

    * Radiation to < 25% of the bone marrow; whole pelvis radiation is excluded.
    * Prior radiotherapy must be completed at least 2 weeks before randomization.
    * Must have recovered from the acute toxic effects of the treatment before randomized.
    * Prior thoracic radiation must be completed 30 days before study enrollment.
    * Irradiated pulmonary lesions cannot be used as target or non-target lesions (and must be excluded) unless there is previous documented progression of these lesions.
    * Palliative extrathoracic radiotherapy can continue, but these lesions must be excluded as target and non-target lesions.
11. Adequate organ function:

    * Bone marrow reserve: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L. Platelets ≥ 100 x 109/L. Hemoglobin ≥ 9 g/dL.
    * Hepatic: Total bilirubin ≤ 1.5 x the upper limit of normal (ULN). Alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT), and lactate dehydrogenase (LDH) and alkaline phosphatase ≤ 2.5 x ULN.
    * Renal: Serum creatinine ≤ 1.5 x ULN, or for participants with serum creatinine > 1.5 ULN, creatinine clearance ≥ 50 mL/min/1.73 m2 (50mL/min/1.73m2 is equivalent to 0.83 mL/s/m2).
12. Participants of childbearing potential:

    * Women who are capable of becoming pregnant must have a negative serum pregnancy test within 1 week prior to exposure to EC20 and within 1 week prior to exposure to treatment with EC145 and/or docetaxel.
    * Women who are capable of becoming pregnant and male participants who are sexually active must practice an effective method of birth control for the duration of their participation in the trial through 3 months following the last dose of EC145 and through 6 months following the last dose of docetaxel.

Exclusion Criteria:

1. Prior therapy with docetaxel, vinorelbine, or vinca-containing compounds.
2. Known hypersensitivity to docetaxel or polysorbate 80.
3. Symptomatic central nervous system (CNS) metastases or metastases that result in midline shift, significant edema.
4. Malignancies other than NSCLC that are expected to alter life expectancy or may interfere with disease assessment. Patients with adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, or low-grade (Gleason score ≤ 6) localized prostate cancer and patients with prior history of malignancy who have been disease free for more than 3 years are eligible.
5. Serious cardiac illness or medical conditions such as unstable angina, pulmonary embolism, or uncontrolled hypertension.
6. Anti-folate therapy such as methotrexate for rheumatoid arthritis.
7. Baseline peripheral neuropathy CTCAE ≥ Grade 2.
8. Pregnant or lactating women.
9. Other concurrent chemotherapy, immunotherapy, radiotherapy, or investigational therapy.
10. Active infections (e.g., hepatitis or HIV carriers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Progression free survival(PFS)based on investigator assessment using RECIST v1.1 | From date of baseline disease assessment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 26 months
  Disease assessment will be conducted via CT/ MRI every 6 weeks while on study. Participants who come off study due to any other reason except progression of disease or death will be followed via CT/ MRI every 6 weeks until disease progression or until start of new therapy.

SECONDARY OUTCOMES:
Compare overall response rate of participants between treatment arms. | up to 26 months
  Analysis will occur when approximately 50% of the PFS events have occurred (for each comparison) and when 94 PFS events have occurred.
Compare disease control rate of participants between treatment arms. | up to 26 months
  Analysis will occur when approximately 50% of the PFS events have occurred (for each comparison) and when 94 PFS events have occurred.
Compare duration of response of participants between treatment arms. | up to 26 months
  Analysis will occur when approximately 50% of the PFS events gave occurred (for each comparison) and when 94 PFS events have occurred.
Compare duration of disease control of participants between treatment arms. | up to 26 months
  Analysis will occur when approximately 50% of the PFS events gave occurred (for each comparison) and when 94 PFS events have occurred.
Compare overall survival of participants between treatment arms. | up to 26 months
  Analysis will occur when approximately 50% of the PFS events gave occurred (for each comparison) and when 94 PFS events have occurred.
Incidence of Adverse Events, Serious Adverse Events, and Deaths. | up to 26 months
  Adverse events (as a measure of safety and tolerability) will be assessed at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Binh Nguyen, MD, PhD, Study Director — Endocyte